CLINICAL TRIAL: NCT07173244
Title: A Real-world Study of Adebrelimab-based Combination Regimens in the Treatment of Advanced Solid Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Tianjin First Central Hospital (Other)
Responsible Party: Principal Investigator, Wei Jiang, Professor, Tianjin First Central Hospital
Other Study IDs: cancer-rws-001
Record Dates: First submitted 2025-08-26; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer; Small Cell Lung Cancer; Gastrointestinal Cancers
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm 1: adebrelimab-based regimen
  Interventions: Drug: Adebrelimab

INTERVENTIONS:
Drug: Adebrelimab — adebrelimab-based regimen

SUMMARY:
This prospective, multicenter, non-interventional, observational, real-world study was designed to evaluate the safety and efficacy of an adebrelimab-based regimen in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This prospective, multicenter, non-interventional, observational, real-world study aims to evaluate the safety and efficacy of adebrelimab in patients with advanced solid tumors. The study is expected to enroll 300 patients with advanced solid tumors. Information on demographics, previous treatment history, adebrelimab-containing treatment regimens, clinical outcomes, and adverse events will be collected for all enrolled patients. Patients must have a clinically confirmed diagnosis of locally advanced, recurrent, or metastatic cancer, including but not limited to non-small cell lung cancer, small cell lung cancer, and gastrointestinal cancers (esophageal, gastric, liver, biliary, pancreatic, and intestinal cancers). Patients had already decided to receive adebrelimab before enrollment. Based on their tumor type, stage, and previous treatment history, they were assigned to one of two cohorts: Cohort 1: First-line treatment with adebrelimab combined with etoposide and carboplatin for extensive-stage small cell lung cancer; Cohort 2: Other solid tumors treated with an adebrelimab-based regimen (excluding central nervous system, urinary, bone, soft tissue sarcomas, and skin tumors such as melanoma). The adebrelimab regimen in Cohort 1 was 1200 mg intravenously infused every 21 days. The adebrelimab regimen in Cohort 2 was based on the instructions. Patients were followed up until loss to follow-up, death, withdrawal of consent, or study termination/closure, whichever occurred first. This study was a non-interventional, real-world study. The diagnosis and treatment process, visits, and examinations were based on routine clinical experience, and no intervention was made on patients' medication choices. The data for this study were primarily sourced from patients' daily diagnosis and treatment records.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and voluntarily enrolled in this study;
2. Histologically or cytologically confirmed extensive-stage small cell lung cancer;
3. Patients with other types of advanced solid tumors confirmed by histology or cytology; patients who, based on currently available data, the investigator believes may benefit from adebrelimab treatment may also be considered for enrollment;
4. Patients in Cohort 1 who experience disease progression and whose second-line treatment options, as assessed by the investigator, include adebrelimab in combination therapy may be enrolled in Cohort 2;
5. Age 18-80 years;
6. Patients deemed by the investigator to be eligible for adebrelimab monotherapy or combination therapy;
7. Female patients of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to the first dose of study drug (Cycle 1, Day 1). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Females and males of childbearing potential must agree to use appropriate contraceptive methods or undergo surgical sterilization during the trial and within 90 days after the last dose of the trial drug.
8. Ability to comply with study and follow-up procedures.

Exclusion Criteria:

1. Women who have been confirmed to be pregnant or breastfeeding;
2. Patients with histologically or cytologically confirmed central nervous system tumors, urinary system tumors, reproductive system tumors, bone tumors, soft tissue sarcomas, melanomas and other skin tumors;
3. Patients with a history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
4. Patients with known allergies to adebrelimab or any of its drugs and excipients;
5. Patients who are deemed by the investigator to be unsuitable for participation in this study in any other circumstances, including but not limited to the following: (1) Patients with autoimmune diseases (AIDs), especially neurological AIDs, or AIDs that are moderate to severe or in active stage and cannot be controlled by immunosuppressants or require high-dose immunosuppressants to control symptoms; (2) Patients with tuberculosis infection, active tuberculosis, and suspected active TB should be examined by chest X-ray, sputum, and clinical symptoms and signs to exclude; (3) The patient has previously received or is about to receive solid organ transplantation or hematopoietic stem cell transplantation; (4) The patient needs to use large doses of antibiotics, glucocorticoids, proton pump inhibitors and other drugs for a long time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced/recurrent or metastatic solid tumors were eligible for adebrelimab-based monotherapy or combination therapy at the investigator's discretion at the time of enrollment. Patients with central nervous system tumors, urinary system tumors, reproductive system tumors, bone tumors, soft tissue sarcomas, melanoma, and other skin tumors were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
The rate of treatment-related adverse reactions(TRAE)/immunotherapy-related adverse reactions/(irAE) and grade ≥ 3 TRAE/irAE | Through study completion, an average of 1 year
  The rate of treatment-related adverse reactions(TRAE)/immunotherapy-related adverse reactions/(irAE) and grade ≥ 3 TRAE/irAE, based on CTAE 5.0

SECONDARY OUTCOMES:
The rate of treatment Mode | Through study completion, an average of 1 year
  The detailed treatment regimen used for enrolled patients
The rate of treatment Mode | Through study completion, an average of 1 year
  The duration of drug treatment (DOT) of eroolled patients
The rate of Treatment efficacy | Through study completion, an average of 1 year
  Statistical analysis of disease-free survival(PFS, median PFS, 1-year PFS rate et.al ) for different treatment regimens
The rate of Treatment efficacy | Through study completion, an average of 1 year
  Statistics of overall survival(OS, median OS, 1-year OS rate et al.) of different treatment regimens
The rate of Treatment efficacy | Through study completion, an average of 1 year
  Statistics on the quality of life of patients with different treatment options, according to Quality of Life Questionnare-Core 30(EORTC QLQ-C30).

IPD SHARING:
Plan to Share IPD: No